CLINICAL TRIAL: NCT01852162
Title: Pharmacodynamic Effects of Dabigatran in Patients With Coronary Artery Disease on Dual Antiplatelet Therapy With Aspirin and Clopidogrel
Brief Title: Pharmacodynamic Effects of Dabigatran in Patients on Dual Antiplatelet Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFJ 2011-112
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; antiplatelet therapy; anticoagulant therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dabigatran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dabigatran (Experimental): Dabigatran 150mg
  Interventions: Drug: Dabigatran
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dabigatran — Dabigatran 150mg
  Other Names: Pradaxa
  Arms: Dabigatran
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
Dual antiplatelet therapy consisting of aspirin and clopidogrel is the cornerstone of treatment for prevention of atherothrombotic events in patients with coronary artery disease (CAD) undergoing percutaneous coronary interventions (PCI). Many patients on dual antiplatelet therapy in this setting may be affected by other thromboembolic conditions, in particular atrial fibrillation, therefore having an indication to also receive oral anticoagulation for stroke prevention. Thus, a considerable percentage of patients are under "triple therapy" which consists of aspirin plus clopidogrel plus an oral anticoagulant. The ever raising population with CAD warranting triple therapy and the growing number of patients being treated with dabigatran underscores the importance of understanding the pharmacodynamic effects of this treatment regimen.

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting of aspirin and clopidogrel is the cornerstone of treatment for prevention of atherothrombotic events in patients with coronary artery disease (CAD) undergoing percutaneous coronary interventions (PCI). Many patients on dual antiplatelet therapy in this setting may be affected by other thromboembolic conditions, in particular atrial fibrillation, therefore having an indication to also receive oral anticoagulation for stroke prevention. Thus, a considerable percentage of patients are under "triple therapy" which consists of aspirin plus clopidogrel plus an oral anticoagulant. Although this combination therapy allows a reduction of atherothrombotic and thromboembolic events, patients on triple therapy are at an increased risk of bleeding complications.

Dabigatran, a synthetic, reversible direct thrombin inhibitor, has been studied as an alternative to warfarin in patients with atrial fibrillation and has been shown to be at least as efficacious with a favorable safety profile. In particular, dabigatran at a dose of 110 mg is associated with rates of stroke and systemic embolism similar to warfarin, with lower rates of major hemorrhage, while a dose of 150 mg is associated with lower thrombotic events with similar rates of bleeding events. These findings have led the Food and Drug Administration (FDA) to approve dabigatran for use in atrial fibrillation patients in December 2011 and this has also been implemented in practice guidelines to be a superior strategy to warfarin. However, the FDA only approved the 150mg formulation.

Dabigatran has high affinity and specificity for its target serine protease thrombin, and one small study shows that dabigatran produced potent inhibition of thrombin-induced platelet aggregation in vitro. However, there are no studies assessing the ex vivo pharmacodynamic effects of dabigatran in patients on dual antiplatelet therapy. The ever raising population with CAD warranting triple therapy and the growing number of patients being treated with dabigatran underscores the importance of understanding the pharmacodynamic effects of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known CAD
* On maintenance treatment with aspirin (81 to 325mg per day) and clopidogrel (75 mg per day) for at least for at least 4-weeks as per standard of care.
* Age between 18 and 80 years old.

Exclusion Criteria:

* Transient ischemic attack or ischemic stroke in the past 6 months.
* Prior hemorrhagic stroke (irrespective of timing).
* Known allergies to dabigatran.
* On treatment with Coumadin derivate or have an indication to be on Coumadin treatment (atrial fibrillation, prosthetic valve, DVT/pulmonary embolism).
* Platelet count <80x106/mL
* Active bleeding or hemodynamic instability.
* Creatinine clearance <30 mL/minute.
* Baseline ALT >2.5 times the upper limit of normal.
* Hemoglobin < 10 gm/dL
* Pregnant females*. *Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, randomized, double-blind, placebo-controlled PD study conducted in patients with CAD on maintenance DAPT with aspirin and clopidogrel. Patients were screened at the Division of Cardiology of the University Of Florida College Of Medicine - Jacksonville from February 2012 to December 2013.
Groups:
- Dabigatran: Patients randomized to the dabigatran arm received dabigatran 150mg twice/daily for 7 (±3) days.
- Placebo: Patients randomized to the placebo arm received matching placebo tablets twice/daily for 7 (±3) days.
Period: Overall Study
Arm/Group | Dabigatran | Placebo
Started | 18 | 17
Completed | 14 | 16
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: Patients were considered for analysis of the PD end points if they completed both visits and had a compliance >80% to study drug, clopidogrel and aspirin. All patients who received any dose of study medication were considered for analysis of safety and any other adverse events.
Groups:
- Dabigatran: Dabigatran 150mg tablets
- Placebo: Placebo tablets
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8) | 59 (9) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: TRAP-induced Platelet Aggregation
Description: TRAP-induced platelet aggregation measured by light transmittance aggregometry (LTA) was similar between groups
Time Frame: 1 week
Population: TRAP-induced platelet aggregation
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 14 | 16
percentage of aggregation | 74 (8) | 77 (6)
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Assuming a 20% relative difference in TRAP induced MPA between dabigatran and placebo with a common standard deviation of 10%, 13 patients with available data needed to be randomized to obtain a 95% power and 2-sided alpha=0.05; Test type: Superiority or Other; p < 0.05, ANCOVA — An analysis of covariance (ANCOVA) method with a general linear model, using the corresponding baseline PD value as a covariate, was used to evaluate the comparisons between dabigatran and placebo at 7 days

2. Secondary Outcome: Platelet Reactivity Measured by LTA
Description: Multiple measures of platelet reactivity evaluating purinergic and non-purinergic signaling pathways were assessed by light transmittance aggregometry (LTA).
Time Frame: 1-week
Population: Platelet aggregation measured by LTA
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 14 | 16
percentage of aggregation
  ADP-induced platelet aggregation | 49.5 (16.6) | 44.6 (15.0)
  Arachidonic acid-induced platelet aggregation | 6.9 (18.2) | 6.0 (1.5)
  Collagen-induced platelet aggregation | 42.6 (22.8) | 34.9 (22.0)

3. Secondary Outcome: Platelet Reactivity Measured by Multiple Electrode Aggregometry.
Description: Multiple measures of platelet reactivity evaluating purinergic and non-purinergic signaling pathways were assessed by multiple electrode aggregometry.
Time Frame: 1-week
Population: Platelet aggregation measured by multiple electrode aggregometry.
Measure: Mean (Standard Deviation); unit: arbitrary aggregation units
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 14 | 16
arbitrary aggregation units
  TRAP-induced platelet aggregation | 1176.4 (274) | 1210.6 (275)
  ADP-induced platelet aggregation | 482.2 (199) | 454.0 (227)
  Arachidonic acid-induced platelet aggregation | 238.9 (88) | 230.1 (115)
  Collagen-induced platelet aggregation | 559.4 (180) | 532.5 (182)

4. Secondary Outcome: Clot Kinetic: Thrombin Activity
Description: Parameters related to thrombin activity and velocity of thrombus generation (reaction time: R; time to maximum rate of thrombus generation: TMRTG) were evaluated by thromboelastography.
Time Frame: 1-week
Population: Clot kinetic assessed by citrated-kaolin thromboelastography
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 14 | 16
minutes
  R | 12.25 (2.6) | 6.76 (1.1)
  TMRTG | 14.32 (3) | 8.4 (1.6)

5. Secondary Outcome: Clot Kinetic: Clot Stength
Description: Clot strength (maximal amplitude:MA) was assessed by thromboelastography.
Time Frame: 1-week
Population: Clot kinetic assessed by citrated-kaolin thromboelastography
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 14 | 16
mm | 63.7 (4.4) | 62.9 (6.7)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Dabigatran | Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran (N=18) | Placebo (N=17)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — One patient in the dabigatran group had a non-ST-segment elevation myocardial infarction during study treatment, which was medically managed and required study drug discontinuation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes